CLINICAL TRIAL: NCT05504291
Title: Intravitreal Melphalan for Intraocular Retinoblastoma
Brief Title: A Study to Give Treatment Inside the Eye to Treat Retinoblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARET2121; NCI-2022-06082 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARET2121 (Other: Children's Oncology Group); ARET2121 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2022-08-04; First posted 2022-08-17 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-04

CONDITIONS: Bilateral Retinoblastoma; Childhood Intraocular Retinoblastoma; Group D Retinoblastoma; Stage I Retinoblastoma; Unilateral Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Specimen Handling; Carboplatin; Etoposide; Magnetic Resonance Spectroscopy; Melphalan; Microscopy, Acoustic; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CVE, melphalan) (Experimental): See Detailed Description
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Procedure: Examination Under Anesthesia; Procedure: Magnetic Resonance Imaging; Drug: Melphalan; Procedure: Ultrasound Biomicroscopy; Drug: Vincristine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo aqueous humor, tissue, and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Procedure: Examination Under Anesthesia — Undergo imaging of the eye during EUA
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Melphalan — Given I-VITRE
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Ultrasound Biomicroscopy — Undergo UBM during EUA
  Other Names: Ultrasound Biomicroscopy (UBM)
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This phase II trial tests the safety and side effects of adding melphalan (by injecting it into the eye) to standard chemotherapy in early treatment of patients with retinoblastoma (RB). RB is a type of cancer that forms in the tissues of the retina (the light-sensitive layers of nerve tissue at the back of the eye). It may be hereditary or nonhereditary (sporadic). RB is considered harder to treat (higher risk) when there are vitreous seeds present. Vitreous seeds are RB tumors in the jelly-like fluid of the eye (called the vitreous humor). The term, risk, refers to the chance of the cancer not responding to treatment or coming back after treatment. Melphalan is in a class of medications called alkylating agents. It may kill cancer cells by damaging their deoxyribonucleic acid (DNA) and stopping them from dividing. Other chemotherapy drugs given during this trial include carboplatin, vincristine, and etoposide. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of cancer cells. Vincristine is in a class of medications called vinca alkaloids. It works by stopping cancer cells from growing and dividing and may kill them. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair and may kill cancer cells. Adding melphalan to standard chemotherapy early in treatment may improve the ability to treat vitreous seeds and may be better than standard chemotherapy alone in treating retinoblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of administering intravitreal melphalan by cycle 6 when given in combination with systemic carboplatin, vincristine, and etoposide (CVE) for the treatment of Group D retinoblastoma with vitreous seeding.

SECONDARY OBJECTIVES:

I. To determine the safety and toxicity profile associated with intravitreal melphalan in combination with systemic CVE for the treatment of Group D retinoblastoma with vitreous seeding.

II. To evaluate the efficacy of intravitreal melphalan in conjunction with systemic chemotherapy in Group D intraocular retinoblastoma with vitreous seeding.

EXPLORATORY OBJECTIVES:

I. To determine if eyes that become eligible for injection at cycle 3 or later would have been eligible for injection at diagnosis by retrospective central review of examination under anesthesia (EUA) and ultrasound biomicroscopy (UBM) images from diagnosis.

II. To validate and standardize the extraction, storage and collection protocols across multiple centers to demonstrate that aqueous humor from eyes undergoing therapy have high enough tumor-derived deoxyribonucleic acid (DNA) concentration for whole genome sequencing and RB1 testing.

III. To explore the relationship between highly-recurrent retinoblastoma (RB) somatic copy number alterations (SCNAs) and ocular salvage as well as tumor fraction (% of tumor DNA) as a marker of minimal residual disease and risk of intraocular disease relapse.

IV. To evaluate the effects of intravitreal melphalan therapy in the histopathology of enucleated eyes for progressive or recalcitrant retinoblastoma while on therapy.

V. To evaluate the long-term visual potential of eyes salvaged using intravitreal therapy.

OUTLINE:

CYCLES 1-2: Patients receive CVE regimen consisting of: carboplatin intravenously (IV) over 15-60 minutes on days 1 and 2 of each cycle, vincristine IV on day 1 of each cycle, and etoposide IV over 90-120 minutes on day 1 and 2 of each cycle. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo ultrasound biomicroscopy (UBM) and imaging of the eye during a procedure called examination under anesthesia (EUA) at baseline and prior to each cycle, and urine sample collection at baseline and on study. NOTE: UBM is completed prior to cycle 1 only.

CYCLES 3+: Patients receive CVE regimen as in cycles 1-2. Patients also undergo EUA prior to each cycle to determine eligibility to receive melphalan. If found eligible, patients receive intravitreal injection of melphalan once between days -14 to 14 of each cycle. Patients who are not eligible for melphalan for any cycle receive CVE only regimen for that cycle. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo urine sample collection at baseline and on study for Cycles 3-6. NOTE: Patients may be eligible to receive additional cycles of melphalan alone (maximum of 6 injections).

Additionally, patients undergo magnetic resonance imaging and may undergo aqueous humor and tissue sample collection throughout the trial.

After completion of study treatment, patients are followed up at 4 weeks, then every 3 months for 1 year, and then every 3-6 months for years 2-5.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be < 18 years of age at enrollment
* Patient must have newly diagnosed intraocular (localized) retinoblastoma and meet one of the following criteria:

  * Unilateral Group D retinoblastoma with vitreous seeding; OR
  * Bilateral retinoblastoma with worst eye Group D, with vitreous seeding present and the contralateral eye is Group A-C; OR
  * Bilateral Group D retinoblastoma with at least one eye with vitreous seeding; OR
  * Bilateral retinoblastoma with one Group D eye with vitreous seeding and one Group E eye where the Group E eye has been enucleated prior to any therapy. Note exclusion for high-risk features
  * Bilateral retinoblastoma with one Group D eye with vitreous seeding and one Group E eye where the Group E eye has not been enucleated prior to any therapy at the discretion of the treating physician. Note exclusion for patients with evidence of metastatic or extra orbital spread
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =<16 years of age
* Peripheral absolute neutrophil count (ANC) >= 750/uL (must be performed within 7 days prior to enrollment unless otherwise indicated)
* Platelet count >= 75,000/uL (transfusion independent) (must be performed within 7 days prior to enrollment)
* A serum creatinine based on age/sex as follows (must be performed within 7 days prior to enrollment; must be repeated prior to the start of protocol therapy if > 7 days have elapsed from their most recent prior assessment):

  * 1 month to < 6 months = 0.4 (male and female)
  * 6 months to < 1 year = 0.5 (male and female)
  * 1 to < 2 years = 0.6 (male and female)
  * 2 to < 6 years = 0.8 (male and female)
  * 6 to < 10 years = 1.0 (male and female)
  * 10 to < 13 years = 1.2 (male and female)
  * 13 to < 16 years = 1.5 (male) and 1.4 (female)
  * >= 16 years = 1.7 (male) and 1.4 (female) OR - a 24-hour urine Creatinine clearance >= 70 mL/min/1.73 m^2 OR - a glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard)
  * Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility

    * For patients < 1 month of age, serum creatinine levels must be < 1.5 x the treating institution's creatinine upper limit of normal (ULN) for patients < 1 month of age or the creatinine clearance or radioisotope GFR must be >= 70 mL/min/1.73 m^2

      * The threshold creatinine values were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Center for Disease Control (CDC)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (must be performed within 7 days prior to enrollment; must be repeated prior to the start of protocol therapy if > 7 days have elapsed from their most recent prior assessment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (must be performed within 7 days prior to enrollment; must be repeated prior to the start of protocol therapy if > 7 days have elapsed from their most recent prior assessment)

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L

Exclusion Criteria:

* Patients with evidence of metastatic or extra-orbital spread
* Patients must not have an invasive infection at time of protocol entry
* Patients must not have had any prior anti-cancer therapy other than cryotherapy and/or laser therapy (green or infrared) to the study eye(s) and non-study eye, including systemic chemotherapy, intra-arterial chemotherapy, radioactive plaque, brachytherapy, or radiation therapy.

  * Note: A study eye is defined as being Group D with vitreous seeding. Patients may have had enucleation of one eye as long as the remaining eye is Group D with vitreous seeds
* Patients with bilateral disease who undergo enucleation of a Group E eye prior to initiation of therapy and show evidence of high-risk histopathology features in the enucleated eye. High-risk histopathology includes choroid involvement >= 3 mm, post lamina optic nerve involvement, full thickness scleral invasion or optic nerve invasion to the cut end
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility success rate of intravitreal melphalan injection in combination with systemic chemotherapy | Up to cycle 6 (1 cycle = 28 days)
  A patient will be considered to have experienced intravitreal injection feasibility success if intravitreal melphalan can be delivered by cycle 6. If the treating physician does not inject because the eye has a full complete response (CR) for vitreous seeds after 2 cycles of systemic chemotherapy, it will be counted as a success in the feasibility analysis. Any feasibility evaluable patient who does not experience feasibility success will be considered a feasibility failure. For a bilateral patient with two Group D eyes with vitreous seeds, he/she will be categorized based on the worse results with the intent of being conservative, i.e., if intravitreal melphalan can be delivered in one eye but not the other by cycle 6 for any reason other than a CR of vitreal seeds, the patient will be deemed as experiencing a failure.

SECONDARY OUTCOMES:
Percentage of patients with grade 3 or higher toxicities | Up to 30 days after last dose of study treatment
  Any eligible patient who receives protocol therapy will be considered as evaluable for toxicity.
Event-free survival (EFS) | Up to 5 years
  Any eligible patient who receives protocol therapy will be considered as evaluable for EFS. Patients who need non-protocol chemotherapy for either the study eye or non-study eye, external beam radiotherapy for either the study eye or non-study eye, or enucleation for the study eye will be considered as having a treatment failure and be considered as experiencing EFS events. The analysis will be conducted per patient level. The EFS along with the 95% confidence intervals will be estimated using the Kaplan-Meier method.

OTHER OUTCOMES:
Retrospective central review of examination under anesthesia and ultrasound biomicroscopy images | Cycle 3 or later(1 cycle = 28 days)
  In order to determine if eyes that become eligible for injection at cycle 3 or later would have been eligible for injection at diagnosis, the retrospective central review on images from diagnosis for eyes that are eligible for injection at cycle 3 or later will be summarized.
Validate and standardize the aqueous humor extraction, storage, and collection protocols across multiple centers | Up to 5 years
  Extract tumor-derived deoxyribonucleic acid (DNA), from aqueous humor, for whole genome sequencing and retinoblastoma (RB)1 testing.
Highly-recurrent RB somatic copy number alterations (SCNAs) tumor fraction | Up to 5 years
  Will explore the relationship between highly-recurrent RB SCNAs and tumor fraction (% of tumor DNA) as a marker of minimal residual disease and risk of intraocular disease relapse.
Tumor fraction | Up to 5 years
  Will explore the relationship between highly-recurrent RB SCNAs and ocular salvage as well as tumor fraction (% of tumor DNA) as a marker of minimal residual disease and risk of intraocular disease relapse.
Proportion of enucleated eyes with particular histopathological characteristics that are known or suspected to affect prognosis adversely | Up to 5 years
  Will be calculated along with the 95% confidence interval. The number of evaluable eyes for this aim will depend on the ocular salvage rate.
Long-term visual potential | Up to 5 years
  Eligible patients who retain the affected eye will be evaluated for visual acuity. The visual acuity will be evaluated prior to cycle 1 and at one year from end of therapy, if age-appropriate. The visual acuity data will be summarized by evaluation time points.

CONTACTS AND LOCATIONS:
Overall Officials: Rachana Shah, Principal Investigator — Children's Oncology Group
Locations (19):
- United States (17):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Perth Children's Hospital, Perth, Western Australia, Australia
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada